CLINICAL TRIAL: NCT03210077
Title: Romanian Entropy Clinical Study Network
Acronym: ROEntropy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Romanian Society of Anesthesia and Intensive Care (Other)
Responsible Party: Principal Investigator, Alexandru Florin Rogobete, MSc, PhDs, Clinical Researcher, Romanian Society of Anesthesia and Intensive Care
Other Study IDs: ROE20171
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: General Anesthetic Drug Adverse Reaction
Keywords: general anesthesia; Entropy; Hypnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Entropy Group: General Anesthesia using Entropy Monitoring
  Interventions: Device: Monitoring
- Control Group: General Anesthesia without Entropy (Control Group)

INTERVENTIONS:
Device: Monitoring — Monitoring
  Groups: Entropy Group

SUMMARY:
The critically ill patient is one of the most complex cases with regard to the optimization of the anesthesia, as well as postoperative management. One of the most important steps in the complex management of such patients is the modulation of anesthesia for every patient needs. We start with the assumptions that the optimization of anesthesia should depend on each patient, being conducted in an individual manner. We also believe that by individualizing the anesthesia by monitoring the entropy it is possible to obtain an appropriate management regarding hemodynamic complications during anesthesia including tachycardia, bradycardia, hypotension and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I, II, III;
* written consent accepted to be enrolled in the study; in polytrauma patients in the operation theatre who are brought directly through the emergency department, written consent is obtained from the relatives, in accordance to the national law number 206, of 2004, for a good and correct scientific research, in the situation where the patient is no capable to sign or give the written consent;

Exclusion Criteria:

* cardiac pacemaker;
* atrial fibrillation at the time of presentation in the operation theatre;
* any subject with epidural catheter, placed pre-operatively;
* allergy to Propofol or another anesthetic drugs;
* pregnancy;
* presence of neuromuscular disease;
* presence of neurologic disease;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who needs general anesthesia and meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of systolic blood pressure baseline | Change from Baseline Systolic Blood Pressure at 10 minutes
  Evaluating the impact of general anesthesia guided with Entropy on the hemodynamic instability in the critically ill patient; hemodynamic instability is represented and characterized by high blood pressure episodes (hypertension), or low blood pressure (hypotension).
Change of heart beat rate baseline | Change from Baseline heart rate at 10 minutes
  Evaluating the impact of general anesthesia guided with Entropy on the heart rate in the critically ill polytrauma patient; cardiac rate instability is represented and characterized by high cardiac rate (tachycardia), or low cardiac rate (bradycardia)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Florin Rogobete, PhDs, Principal Investigator — Romanian Society of Anesthesia and Intensive Care; Dorel Sandesc, Prof, Study Chair — Romanian Society of Anesthesia and Intensive Care; Ovidiu Bedreag, Assoc Prof, Study Director — Romanian Society of Anesthesia and Intensive Care
Locations (1):
- Romanian Society of Anesthesia and Intensive Care, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No